CLINICAL TRIAL: NCT06411314
Title: Efficacy and Safety of Vaginal Suppositories Containing Combination of Natamycin and Lactulose in Treatment of Vulvovaginal Candidiasis: International, Randomized, Controlled, Superiority Clinical Trial
Brief Title: Efficacy and Safety of Natamycin and Lactulose Vaginal Suppositories in Treatment of Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avva Rus, JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/21-AVVA RUS
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Vulvovaginal Candidiasis, Genital
Keywords: vulvovaginal candidiasis; itching; Natamycin; Lactulose
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Pruritus | interventions — Natamycin; Lactulose; Suppositories

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Natamycin + Lactulose 100 mg + 300 mg vaginal suppositories (Experimental)
  Interventions: Combination Product: Natamycin + Lactulose 100 mg + 300 mg vaginal suppositories
- Lactulose 300 mg vaginal suppositories (Active Comparator)
  Interventions: Drug: Lactulose 300 mg vaginal suppositories
- Pimafucin® (natamycin) 100 mg vaginal suppositories (Active Comparator)
  Interventions: Drug: Pimafucin® (natamycin) 100 mg vaginal suppositories

INTERVENTIONS:
Combination Product: Natamycin + Lactulose 100 mg + 300 mg vaginal suppositories — 1 suppository once daily at bedtime for 6 days
  Arms: Natamycin + Lactulose 100 mg + 300 mg vaginal suppositories
Drug: Lactulose 300 mg vaginal suppositories — 1 suppository once daily at bedtime for 6 days
  Arms: Lactulose 300 mg vaginal suppositories
Drug: Pimafucin® (natamycin) 100 mg vaginal suppositories — 1 suppository once daily at bedtime for 6 days
  Arms: Pimafucin® (natamycin) 100 mg vaginal suppositories

SUMMARY:
The purpose is to study superior efficacy of combination of Natamycin and Lactulose (Natamycin 100 mg + Lactulose 300 mg vaginal suppositories) compared to Pimafucin (Natamycin 100 mg vaginal suppositories), or Lactulose 300 mg vaginal suppositories. The second objective of the study was to investigate the safety of the combination suppositories in the treatment of vulvovaginal candidiasis in non-pregnant adult females.

ELIGIBILITY:
Inclusion Criteria:

* two or more of the following signs and symptoms of vulvovaginal candidiasis: white or yellowish-white curd-like, thick or creamy vaginal discharge; vulvar itching, burning and pain; anogenital itching and burning; discomfort in the vulva; itching, burning, painful urination (dysuria);
* yeast cells in the vaginal swab specimen;
* vaginal pH ≤ 4.5.

Exclusion Criteria:

* a clinical and laboratory diagnosis of bacterial vaginosis; vulvovaginitis caused by specific pathogens such as Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhoeae; chronic inflammatory, atrophic, or oncologic diseases of the female genital tract; previous surgery on external or internal genitalia within 6 months; childbirth and abortion within 6 months.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of patients who achieved a clinical response (recovery) at Visit 2 | 7 days
  The clinical response was considered as the absence of significant signs and symptoms of VVC (white or yellowish-white curd-like, thick, or creamy vaginal discharge; vulvar itching, burning and pain; anogenital itching and burning; discomfort in the vulva; itching, burning, painful urination [dysuria])

SECONDARY OUTCOMES:
Proportion (%) of patients with the clinical response at Visit 3 | 24 days
  The clinical response was considered as the absence of significant signs and symptoms of VVC (white or yellowish-white curd-like, thick, or creamy vaginal discharge; vulvar itching, burning and pain; anogenital itching and burning; discomfort in the vulva; itching, burning, painful urination [dysuria])
Proportion (%) of patients with microscopic recovery (absence of Candida spp. at Visits 2 and 3 | 24 days
  The vaginal culture test for Candida spp. was used for the microscopic assessment
Proportion of patients with overall (clinical and microscopic) recovery at Visits 2 and 3 | 24 days
  The vaginal culture test was used for the microscopic assessment
Patient's efficacy assessment by the 5-point scale at Visits 2, 3 | 24 days
  The patient completed a questionnaire in the presence of the investigating physician as part of the efficacy assessment. The questionnaire contained closed-ended responses ranging from 1 point (no clinical symptoms) to 5 points (severe clinical symptoms)
Microscopic change in lactobacilli count in vaginal specimens at Visits 2 and 3 compared to baseline (Visit 0) | 24 days
  Microscopic change in lactobacilli count in vaginal specimens at Visits 2 and 3
Incidence of adverse events | 24 days
  incidence of any adverse events, an incidence of serious adverse events (SAEs), an incidence of AEs and SAEs probably related (in the investigator's opinion) with the study drug at the study dose, and an incidence of AEs and SAEs that led to study drug discontinuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Reproductive Medicine and Surgery at the A.I. Evdokimov Moscow State Medical and Dental University, Moscow, Russia

REFERENCES:
- [Derived] Volkova ON, Amel'chenko EV, Makeeva OV, Tolmachev SA, Lesovaya EA, Zacharia LC, Dikovskiy AV. Efficacy and safety of vaginal suppositories containing combination of Natamycin and Lactulose in treatment of vulvovaginal candidiasis: international, randomized, controlled, superiority clinical trial (combination of Natamycin and Lactulose for treatment of vulvovaginal candidiasis). BMC Womens Health. 2025 Feb 20;25(1):77. doi: 10.1186/s12905-025-03616-3. PMID 39979898